CLINICAL TRIAL: NCT03632941
Title: A Phase II Randomized Study to Evaluate the Immunologic and Antitumor Activity of Concurrent VRP-HER2 Vaccination and Pembrolizumab for Patients With Advanced HER2-overexpressing Breast Cancer
Brief Title: A Study to Evaluate Concurrent VRP-HER2 Vaccination and Pembrolizumab for Patients With Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Lyerly (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Herbert Lyerly, Principal Investigator, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100093
Record Dates: First submitted 2018-08-09; First posted 2018-08-16 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; HER2+ Breast Cancer
Keywords: Cancer; Immunotherapy; PD-1 Antibody; HER2; T cell
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VRP-HER2 Vaccine (Active Comparator): VRP-HER2 Vaccine 4 x 10EE8 IU given as a single injection every 2 weeks for 3 injections total (Cycle 1: Day 1 and Day 15 Cycle 2: Day 8)
  Interventions: Biological: VRP-HER2
- Pembrolizumab (Active Comparator): 5 administrations of Pembrolizumab 200 mg every 3 weeks for 5 total IV infusions (Day 1 of each 3 week cycle x 5 cycles)
  Interventions: Biological: Pembrolizumab
- VRP-HER2 Vaccine + Pembrolizumab (Experimental): VRP-HER2 Vaccine 4 x 10EE8 IU given as a single injection every 2 weeks for 3 injections total (Cycle 1: Day 1 and Day 15 Cycle 2: Day 8)+ 5 administrations of Pembrolizumab 200 mg every 3 weeks for 5 total IV infusions (Day 1 of each 3 week cycle x 5 cycles)
  Interventions: Biological: VRP-HER2; Biological: Pembrolizumab

INTERVENTIONS:
Biological: VRP-HER2 — VRP (alphavirus-like replicon particles) containing self amplifying replicon RNA for HER2
  Other Names: AVX901
  Arms: VRP-HER2 Vaccine; VRP-HER2 Vaccine + Pembrolizumab
Biological: Pembrolizumab — A humanized antibody specific for the programmed cell death 1 (PD-1) receptor.
  Other Names: Keytruda
  Arms: Pembrolizumab; VRP-HER2 Vaccine + Pembrolizumab

SUMMARY:
In this phase II study, participants will receive the VRP-HER2 immunizations plus pembrolizumab. Subjects will be randomized into 3 arms. They will undergo a biopsy of their tumor and peripheral blood draw for immune cell analyses and be assigned to the applicable arm of the study. Arm A will consist of the the VRP-HER2 immunizations; Arm B will consist of pembrolizumab; Arm C will consist of the VRP-HER2 immunizations plus pembrolizumab.

DETAILED DESCRIPTION:
The primary objective of this phase II study is to determine whether pembrolizumab increases the tumor infiltrating and peripheral blood immune response to the VRP-HER2 vaccine. The investigators hypothesize that HER2 specific T cell responses and anti-tumor immunity induced with HER2 vaccination will be augmented by concurrent anti-PD-1 antibody therapy.

The investigators will additionally determine whether the administration of pembrolizumab is safe in patients with recurrent or metastatic HER2+ cancers who are receiving the anti-HER2 vaccine VRP-HER2.

Participants will be randomized 1:1:1 into 3 arms (n=12 per arm). Subjects with metastatic HER2 overexpressing breast cancer receiving trastuzumab and pertuzumab will continue these antibodies. They will undergo a biopsy of their tumor and peripheral blood draw for immune cell analyses and be assigned to the applicable arm of the study. Arm A will consist of the the VRP-HER2 immunizations; Arm B will consist of pembrolizumab; Arm C will consist of the VRP-HER2 immunizations plus pembrolizumab. Tumor biopsies and peripheral blood draws will be performed following the course of immunizations.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone treatment with trastuzumab plus pertuzumab for at least 3 weeks prior to initiation on this study.
* Be willing and able to provide written informed consent/assent for the trial.
* Resolution of all toxic side effects of prior chemotherapy, radiotherapy or surgical procedures to NCI CTCAE (version 4.03) Grade ≤ 1 (with the exception of grade 2 alopecia, grade 2 neuropathy and grade 2 fatigue);
* Be >=18 years of age on day of signing informed consent.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.. Subjects for whom newly-obtained samples cannot be provided may submit an archived specimen only upon agreement from the Sponsor.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Normal cardiac function defined as either a MUGA or ECHO with LVEF in normal institutional range.
* Demonstrate adequate organ function as defined below:

System Laboratory Value Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency

Serum creatinine OR Measured or calculated creatinine clearance

* 1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT)

* 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

* Male subjects of childbearing potential must agree to use an adequate method of contraception.
* Ability to return to Duke University Medical Center for adequate follow-up as required by this protocol.

Exclusion Criteria:

* Patients in this study, may not receive cytotoxic chemotherapy, anti-estrogen therapy, targeted small molecule therapy, or radiation therapy in the 3 weeks before the first infusion of Pembrolizumab, during the injection period for VRP-HER2 and infusion period for Pembrolizumab or for at least 2 weeks after booster immunization with VRP-HER2 (Arm 1) or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Patients may have received prior radiation including for brain metastases.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 3 months prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Prior history of autoimmune thyroiditis or vitiligo is permitted.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has history of (non-infectious) pneumonitis that required steroids or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy or systemic use of antimicrobials within 72 hours prior to the first study treatment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA is detected).
* Has received a live vaccine within 30 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crosby EJ, Acharya CR, Haddad AF, Rabiola CA, Lei G, Wei JP, Yang XY, Wang T, Liu CX, Wagner KU, Muller WJ, Chodosh LA, Broadwater G, Hyslop T, Shepherd JH, Hollern DP, He X, Perou CM, Chai S, Ashby BK, Vincent BG, Snyder JC, Force J, Morse MA, Lyerly HK, Hartman ZC. Stimulation of Oncogene-Specific Tumor-Infiltrating T Cells through Combined Vaccine and alphaPD-1 Enable Sustained Antitumor Responses against Established HER2 Breast Cancer. Clin Cancer Res. 2020 Sep 1;26(17):4670-4681. doi: 10.1158/1078-0432.CCR-20-0389. Epub 2020 Jul 30. PMID 32732224

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VRP-HER2 Vaccine | Pembrolizumab | VRP-HER2 Vaccine + Pembrolizumab
Started | 1 | 2 | 5
Completed | 1 | 2 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VRP-HER2 Vaccine | Pembrolizumab | VRP-HER2 Vaccine + Pembrolizumab | Total
Number analyzed (Participants) | 1 | 2 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (NA) — No SD available as there was only one participant in this group. | 52.0 (12.7) | 63.8 (9.5) | 57.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 8
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 1 | 2 | 3 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Positive T Cell Response Based on ELISpot Results
Description: The enzyme-linked immunosorbent spot (ELISpot) assay is a quantitative method that measures the frequency of cytokine secretion in a single cell.
Time Frame: up to approximately 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VRP-HER2 Vaccine | Pembrolizumab | VRP-HER2 Vaccine + Pembrolizumab
Number analyzed (Participants) | 1 | 2 | 5
Participants | 1 | 1 | 3

2. Secondary Outcome: Number of Participants With a Severe Adverse Event as Assessed by CTCAE v5.0
Description: Adverse events are graded on a scale from 1 to 5. Grade 1 adverse events are mild and generally not bothersome. Grade 2 events are bothersome and may interfere with doing some activities but are not dangerous. Grade 3 events are serious and interfere with a person's ability to do basic things like eat or get dressed. Grade 3 events may also require medical intervention. Grade 4 events are usually severe enough to require hospitalization. Grade 5 events are fatal. Reported here is the number of participants with a grade 3 adverse event.
Time Frame: up to approximately 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | VRP-HER2 Vaccine | Pembrolizumab | VRP-HER2 Vaccine + Pembrolizumab
Number analyzed (Participants) | 1 | 2 | 5
Participants | 0 | 0 | 1

3. Other Pre Specified Outcome: Number of Participants With Stable Disease as Overall Response Based on RECIST 1.1 Criteria
Description: RECIST (Response Evaluation Criteria in Solid Tumors) defines Stable Disease as neither partial response (>30% decrease in the sum of diameters of target lesions) or progressive disease (<20% decrease in the sum of diameters of target lesions).
Time Frame: up to approximately 15 weeks
Population: Data not collected on 1 participant in the VRP-HER2 Vaccine group and 1 participant in the Pembrolizumab group.
Measure: Count of Participants; unit: Participants
Arm/Group | VRP-HER2 Vaccine | Pembrolizumab | VRP-HER2 Vaccine + Pembrolizumab
Number analyzed (Participants) | 1 | 1 | 4
Participants | 1 | 1 | 4

ADVERSE EVENTS:
Time Frame: Up to approximately 15 weeks
Arm/Group | VRP-HER2 Vaccine | Pembrolizumab | VRP-HER2 Vaccine + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 1/5
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VRP-HER2 Vaccine (N=1) | Pembrolizumab (N=2) | VRP-HER2 Vaccine + Pembrolizumab (N=5)
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Creatinine increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VRP-HER2 Vaccine (N=1) | Pembrolizumab (N=2) | VRP-HER2 Vaccine + Pembrolizumab (N=5)
Plantar Warts (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Localized edema (General disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Edema face (General disorders) | 0 | 1 | 0
Exacerbation of Psoriasis- bilateral hands (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2
Hot flashes (Vascular disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 3
Fatigue (General disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03632941/Prot_SAP_000.pdf